CLINICAL TRIAL: NCT06458543
Title: Efficacy of Bovhyaluronidase Azoximer on Biofilms Destruction in the Urogenital Tract of the Patients With Reccurent Bacterial Vaginosis.
Brief Title: Optimization of Bacterial Vaginosis Treatment in Women of Reproductive Age
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Longidaza IMSechenovMMA; NCT06453200 (obsolete NCT alias)
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-06

CONDITIONS: Bacterial Vaginosis
Keywords: Bacterial Vaginosis; biofilms; bovhyaluronidase azoximer; treatment
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Longidaza; Metronidazole; Benchmarking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group includes 50 women of reproductive age (18 - 45 years old) with an established diagnosis of bacterial vaginosis.
  Participants in the experimental group will be given the drug Bovgialuronidase azoximer and Metronidazole.
  Bovhyaluronidase azoximer, vaginal suppositories 3000 IU, 1 suppository vaginally every other day, course of 10 days Metronidazole, tablets 500 mg, 1 tablet 2 times a day, orally, course 7 days
  Interventions: Drug: Longidaza; Drug: Metronidazole 500 mg
- Control (Active Comparator): The control group includes 50 women of reproductive age (18 - 45 years old) with an established diagnosis of bacterial vaginosis.
  Metronidazole, tablets 500 mg, 1 tablet 2 times a day, orally, course 7 days
  Interventions: Drug: Metronidazole 500 mg

INTERVENTIONS:
Drug: Longidaza — Bovhyaluronidase azoximer, vaginal suppositories 3000 IU, 1 suppository vaginally every other day, course of 10 days
  Other Names: Bovhyaluronidase azoximer
  Arms: Experimental
Drug: Metronidazole 500 mg — Metronidazole, tablets 500 mg, 1 tablet 2 times a day, orally, course 7 days
  Other Names: Metronidazol

SUMMARY:
The purpose of this clinical trial is to study the efficacy of bovgialuronidase azoximere in the treatment and duration of recurrence-free course of bacterial vaginosis in women of reproductive age. The main questions it aims to answer are:

* Is bovgialuronidase azoximer able to destroy G. vaginalis associated biofilms of the vaginal epithelium
* use of bovgialuronidase azoximer together with Metronidazole increases the effectiveness of treatment of bacterial vaginosis.
* use of azoximers bovgialuronidase together with Metronidazole increases the duration of relapse-free course of bacterial vaginosis.

Participants in the experimental and control group will be:

* Amsel criteria assessment
* Colpotest-PH (vaginal acidity)
* aminotest with 10% KOH solution ("fish odor")
* microscopic examination of vaginal discharge
* Bacteriologic culture of vaginal discharge
* Polymerase chain reaction of epithelial cell scrapings from the vagina
* electron microscopy of vaginal epithelial cell scrapings

Participants in the main group will be given the drug Bovgialuronidase azoximer and Metronidazole.

Participants in the control group: Metronidazole.

Researchers will compare the experimental and control groups to see if there are differences after treatment in biofilm structure, treatment efficacy, and duration of recurrence-free survival.

DETAILED DESCRIPTION:
Bacterial vaginosis is characterized by a decrease in the number of lactobacilli and the dominance of opportunistic anaerobic flora (primarily G.vaginalis, to a lesser extent Atopobium vaginae, Peptostreptococcus, Clostridiales spp., Prevotella spp., etc.). Modern ideas of the pathogenesis of bacterial vaginosis consist in the formation of polymicrobial biofilms on the surface of the mucosa of the vaginal epithelium. Biofilms are a community of microorganisms of one or more species attached to the surface of a polymeric matrix. Biofilms are formed predominantly by G.vaginalis and to a lesser extent by other pathogens associated with bacterial vaginosis (Atopobium vaginae, Peptostreptococcus, Clostridiales spp., Prevotella spp., etc.). Biofilm-associated bacterial vaginosis is characterized by increased resistance to pathogenetic therapy, the ability to evade defense mechanisms and prolonged persistence in the vaginal environment. These features of pathogenesis cause a high rate of recurrences and chronic course of bacterial vaginosis.

Thus, it is relevant to study in vivo the role of drug action on biofilms to destroy them in order to increase the effectiveness of antibacterial therapy and reduce the frequency of recurrences of bacterial vaginosis.

The standard and approved by the Ministry of Health of the Russian Federation method of treatment of bacterial vaginosis is Metronidazole.

The aim of this clinical trial is to investigate the efficacy of combination therapy with metronidazole and azoximera bovgialuronidase in the treatment and duration of relapse-free course of bacterial vaginosis in women of reproductive age compared with metronidazole monotherapy.

The main questions it aims to answer are:

* Is bovgialuronidase azoximer able to destroy G. vaginalis associated biofilms of the vaginal epithelium
* use of bovgialuronidase azoximer together with Metronidazole increases the effectiveness of treatment of bacterial vaginosis.
* use of azoximers bovgialuronidase together with Metronidazole increases the duration of relapse-free course of bacterial vaginosis.

Participants in the experimental and control group will be:

* Amsel criteria assessment
* Colpotest-PH (vaginal acidity)
* aminotest with 10% KOH solution ("fish odor")
* microscopic examination of vaginal discharge
* Bacteriologic culture of vaginal discharge
* Polymerase chain reaction of epithelial cell scrapings from the vagina
* electron microscopy of vaginal epithelial cell scrapings

Main group - patients with bacterial vaginosis receiving pathogenetic antibacterial therapy (Metronidazole) in combination with Bovgialuronidase azoximer.

Control group - patients with bacterial vaginosis receiving pathogenetic antibacterial therapy (Metronidazole) without Bovgialuronidase azoximer.

Researchers will compare the experimental and control groups to see if there are differences after treatment in biofilm structure, treatment efficacy, and duration of recurrence-free survival.

ELIGIBILITY:
Inclusion Criteria:

* The written informed consent of the patient to participate in the study;
* Age (18 - 45 years old);
* The established diagnosis of Bacterial vaginosis;
* Absence of pregnancy and lactation.

Exclusion Criteria:

* Refusal of the patient from further participation in the study;
* Lack of patient adherence to treatment;
* The occurrence of conditions and diseases related to the list of contraindications to the use of the studied drug during the study.
* The presence of Neisseria gonorrhoeae, Trichomonas vaginalis, confirmed by laboratory;
* The presence of contraindications to the use of the studied drug according to the instructions for the drug.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in the number of relapses of bacterial vaginosis | 6 months after treatment
  Evaluated by clinical data (using Amsel criteria) and laboratory (microscopic examination - identification of "key cells")
  The Amsel criteria include 4 parameters, each of which is scored as one point:
  * gray/white/grayish-white vaginal discharge
  * Vaginal acidity pH greater than 4.5 (colpotest pH)
  * aminotest with 10% solution of potassium hydroxide KOH (appearance of "fishy", "rotten" odor)
  * Presence of "key cell" in microscopic examination of vaginal discharge
  The presence of 3 or more of the 4 criteria speaks in favor of the diagnosis of "bacterial vaginosis" 2 and less points - absence of "bacterial vaginosis"

SECONDARY OUTCOMES:
changes in biofilm structure according to electron microscopy data | 21 days after treatment
  Biofilms are a cooperation of microorganisms of one or more species that are incorporated into a polymeric matrix consisting of proteins, polysaccharides and nucleic acids. Electron microscopy allows to evaluate the structure of the biofilm, to distinguish between lactobacilli and anaerobes (G. vaginalis, Atopobium vaginae, Peptostreptococcus, Clostridiales spp., Prevotella spp., etc.). The destructive effect of azoximers bovgialuronidase on biofilms leads to disruption of biofilm structure: formation of holes in its structure, reduction of its size (volume), release of bacteria from the biofilm structure. Metronidazole has a bactericidal effect on G. vaginalis, Atopobium vaginae, Peptostreptococcus, Clostridiales spp., Prevotella spp., etc., which is expressed in the reduction of CFU/ml.
decrease in the severity of characteristic complaints in female patients with BV | 21 days after treatment
  The main complaints that patients with bacterial vaginosis present with are: vaginal discharge and unpleasant odor of vaginal discharge.
  The Amsel criteria are used to objectively assess these complaints
  The Amsel criteria include 4 parameters, each of which is scored as one point:
  * gray/white/grayish-white vaginal discharge
  * Vaginal acidity pH greater than 4.5 (colpotest pH)
  * aminotest with 10% solution of potassium hydroxide KOH (appearance of "fishy", "rotten" odor)
  * Presence of "key cell" in microscopic examination of vaginal discharge
  The presence of 3 or more of the 4 criteria speaks in favor of the diagnosis of "bacterial vaginosis" 2 and less points - absence of "bacterial vaginosis"
  After treatment the patient is expected to have no characteristic complaints
Decreased vaginal acidity | 21 days after treatment
  Normally, the acidity of the vagina is 4.5 or less (рН=4,5 оr less), meaning the vagina has an acidic environment.
  The pH is measured with the Kolpotest-PH rapid test. After applying vaginal discharge to the indicator screen of the test strip, it is colored. The color obtained is compared with the indicator scale placed on the Colpotest-pH jar. If the pH is 4.5 or less, it is normal.
  A pH result greater than 4.5 favors a diagnosis of bacterial vaginosis After treatment is expected to normalize vaginal acidity (pH = 4.5 or less)
Normalization of the composition of the microflora of the urogenital tract | 21 days after treatment
  Normally, the vagina of women of reproductive age is dominated by Lactobacilli (80-100%). A decrease in lactobacilli or their absence leads to the dominance of opportunistic microorganisms (e.g., G.vaginalis, Atopobium vaginae, Peptostreptococcus, Clostridiales spp., Prevotella spp., etc.), which causes the appearance of complaints characteristic of bacterial vaginosis (vaginal discharge, unpleasant odor of vaginal discharge, itching, burning).
  Microbiome is assessed by polymer chain reaction (Femoflor-16), which allows not only qualitative but also quantitative assessment of the composition of the vaginal microbiome.
  After treatment, the number of opportunistic anaerobes is expected to decrease and the number of lactobacilli is expected to be dominant

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Spivak, MD,Prof., Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University); Kseniya Rossolovskaya, Study Director — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (2):
- Russia (2):
  - LLC "Family polyclinic No. 4" Korolev, Korolyov
  - I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow

IPD SHARING:
Plan to Share IPD: No